CLINICAL TRIAL: NCT05196841
Title: The Effect of Fatima Ana's Hand (Anastatica Hierochuntica) on Birth Pain and Duration: A Randomized Controlled Study
Brief Title: The Effect of Fatima Ana's Hand on Birth Pain and Duration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KaratayUNI
Record Dates: First submitted 2021-11-27; First posted 2022-01-19 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2021-11

CONDITIONS: Labor Pain; Labor Long
Keywords: Labor pain; Labor duration; Midwife; Anastatica Hierochuntica
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Anastatica Hierochuntica
  Interventions: Behavioral: Anastatica Hierochuntica
- Control group (No Intervention): routine care

INTERVENTIONS:
Behavioral: Anastatica Hierochuntica — During the sampling process, the researcher inquired through women who apply for pregnancy follow-up and contacted the mothers who had some inclusion criteria. Also, the researcher outlined the research plan and objectives. The participants were assessed based on the eligibility criteria and, if they were eligible and willing to participate in the study.
  Arms: Experimental group

SUMMARY:
Research Question: Does the Anastatica Hierochuntica have an effect on labor pain and duration? Methods: This study was planned as a a double blind randomized controlled experimental study. The study was conducted with 60 pregnant women who were randomized between February 2019 and November 2020 at a university and private hospital located in Anatolia, Turkey.

DETAILED DESCRIPTION:
Complementary treatment methods during the birth process are supportive therapies. It is applied to meet the physical and psychological care needs, to help cope with pain during childbirth, to increase the quality of life of pregnant women. Mind-body methods, alternative medical methods, biological-based treatment methods, manipulative and body-based methods, and energy therapy methods are used as complementary treatment methods in labor. The focus applied within the scope of mind-body methods is based on the principle of revealing the mental skill that improve bodily functions. One of the methods applied in this direction is Anastatica Hierochuntica.

Anastatika Hierochuntica is a herbaceous plant that can live 1000-2000 years, with dry leaves resembling a fist-closed hand in which it stores its seeds. Known as "Fatma Ana Eli" or "Meryem Ana Eli". This dry ball-shaped plant in the deserts of Namibia comes alive in the rain and turns to green color by opening the folds. After the rain, the leaves of the plant, which stores some water to pass through a new drought period, close again and take a dry appearance.

The plant Anastatica Hierochuntica is known to have a facilitating effect on labor and is frequently used for this purpose during labor. During childbirth, the Anastatica Hierochuntica plant is dropped into a bowl of water. It is believed that as the plant opens, labor will be easier, and the baby will flow like water.

Despite its frequent use, when the literature is examined, no studies hasve been found on the effect of Anastatica Hierochuntica on birth. For this reason, the study was conducted to evaluate the effect of Anastatica Hierochuntica on labor pain and duration.

ELIGIBILITY:
Inclusion Criteria:

* Having a singleton pregnancy at 38-42 weeks,
* Pregnant women who had spontaneous labor,
* Pregnant women with a healthy fetus,
* Pregnant women without any complications that may cause dystocia during labor,
* Pregnant women who did not receive analgesia and anesthesia during the first phase of labor,
* Planned vaginal delivery, pregnant women who volunteered to participate in the research

Exclusion Criteria:

pregnant women with high-risk pregnancies, Planned caesarean delivery, pregnant women with chronic diseases

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Severity of labor pain | 12 hours
  The primary outcomes included the severity of labor pain that was measured by VAS

SECONDARY OUTCOMES:
Duration of the active phase of labor | 12 hours
  The secondary outcomes included the duration of the active phase of labor and the second stage of delivery. The length of delivery stages was recorded in the partograph chart during labor and childbirth by the researcher.

CONTACTS AND LOCATIONS:
Overall Officials: Hediye KARAKOC, PhD, Principal Investigator — Karatay University
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)